CLINICAL TRIAL: NCT05046041
Title: A Study of Acceptability and Feasibility of an Outpatient "Day Procedure" for Medical Abortion at 13-18 Weeks Gestation in Two Public Sector Hospitals in Nepal
Brief Title: Assessing Outpatient 'Day Procedure' for Second-trimester Medical Abortion at Two Public Sector Hospitals in Nepal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: KIST Medical College and Teaching Hospital (Unknown); Center for Research on Environment, Health and Population Activities (Other); Bharatpur Eye Hospital (Other); Lumbini Provincial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1051
Record Dates: First submitted 2021-07-22; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Abortion in Second Trimester
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mifepristone + Misoprostol (Experimental): 200mg mifepristone followed 24-48 h later with 400mcg misoprostol (repeat Q3)
  Interventions: Drug: Mifepristone + Misoprostol

INTERVENTIONS:
Drug: Mifepristone + Misoprostol — A single 200 mg mifepristone (one tablet) to be taken orally either at home or at the hospital, followed approximately 24 - 48 hours later with administration of 400 mcg misoprostol. Repeat doses of 400 mcg (two tablets) of misoprostol will be administered buccally (buccal) every three hours until the abortion is achieved.

SUMMARY:
This study seeks to evaluate the safety, acceptability and feasibility of an outpatient "day procedure" for medical abortion at 13-18 weeks gestation in two public sector facilities. It also seeks to document the roles of health workers in providing services related to later abortion care and to document the costs of this day procedure to the health system.

ELIGIBILITY:
Inclusion Criteria:

1. Have an ongoing pregnancy of 13-18 weeks gestation
2. Meet legal criteria to obtain abortion at 13-18 weeks gestation (Legal criteria include pregnancy resulting from rape or incest, fetal malformation and/or if the pregnancy affects the physical or mental health of the woman)
3. Have access to a phone where she can be reached at the 2-week follow up or willing to return to the clinic for an in-person interview with the research assistant
4. Be willing to follow study procedures

Exclusion Criteria:

1. Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
2. Any contraindications to vaginal delivery
3. More than one prior cesarean delivery
4. Living more than 2 hours away from the hospital

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with method success on the same day as misoprostol initiation. | 0 - 48 hours after first dose of mifepristone
  Success is defined as expelling fetus and placenta without surgical intervention and return home on the same day

SECONDARY OUTCOMES:
Average induction-to-abortion interval | 0 - 48 hours after first misoprostol dose
  Time interval from administration of the first misoprostol dose until expulsion of both fetus and placenta
Average number of total doses of misoprostol | 0 - 48 hours after first misoprostol dose
  Total misoprostol doses administered from induction to delivery of placenta.
Frequency of adverse events | 0-2 weeks after initial visit
  Adverse events include extramural delivery, hemorrhage requiring transfusion, infection, uterine rupture, or prolonged hospitalization, any complications (immediate and delayed)
Description of tasks performed by different cadres of study staff | 0 - 72 hours after receipt of mifepristone
  Tasks evaluated include counseling, monitoring vital signs, administering drugs, monitoring woman's condition, post-abortion contraception, managing discharge
Average total hospital admission time | Within 0 - 48 hours after the second dose of misoprostol
  Total hospital admission time, including: 1) total admission time during treatment with misoprostol and abortion recovery 2) Additional hospital time required for the evaluation and management of complications
Average pain scores | 0 - 48 hours after first dose of misoprostol
  Severity incidence based on a 0-10 point pain scale
Frequency of individual side effects experienced by participants | 0 - 48 hours after first dose of misoprostol
  Side effects evaluated include diarrhea, nausea, vomiting, fever, chills
Proportion of reported complications | 0-2 weeks after initial visit
  Participants who returned to a health facility for evaluation and management of complications within 2 weeks of taking mifepristone
Proportion of satisfied participants | 2 weeks after initial visit
  Participants who report high satisfaction with service

CONTACTS AND LOCATIONS:
Overall Officials: Inga Platais, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, Principal Investigator — Gynuity Health Projects; Anand Tamang, Principal Investigator — CREHPA; Sajan K.C, MD, Principal Investigator — Bharatpur Eye Hospital; Shreedhar Acharya, MD, Principal Investigator — Lumbini Provincial Hospital
Locations (2):
- Nepal (2):
  - Bharatpur Hospital, Bharatpur
  - Lumbini Provincial Hospital, Butwāl